CLINICAL TRIAL: NCT01613105
Title: Prospecitve, Non Interventional, Non Controlled, Post Marketing Survelliance Study to Evaluate Efficacy, Safety, Tolerability of Glucobay on Top of Sulfonylurea Under Daily Life Treatment Conditions
Brief Title: Diabetes Treatment With Glucobay in Combination With Sulfonylurea
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Pharmaceuticals Pvt Ltd
Other Study IDs: 13927; GB0712IN (Other: company internal)
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Type-2; Acarbose; Drug Therapy; Combination
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Acarbose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Acarbose (Precose/Glucobay, BAYG5421)

INTERVENTIONS:
Drug: Acarbose (Precose/Glucobay, BAYG5421) — Oral Glucobay 25 titrated to Glucobay 50 upto three times a day with meals or as per investigators descretion.

SUMMARY:
In this prospective, non interventional, observational Post Marketing Survelliance study data are obtained on the efficacy, safety and tolerability of Glucobay treatment on top of sulfonylurea under daily life treatment conditions.Specifically investigated is the influence of Glucobay on Post Prandial Blood Glucose and HbA1c as well as on pateint's weight when added to an already existing sulfonylurea therapy.The study is planned to carried out in 25000 - 30000 patients from 200 trial sites in India.The Post Marketing Survelliance study will be performed with commercially available medication prescribed within regular practice of the physician. No other examination will be performed than would be done without Post Marketing Survelliance study.

ELIGIBILITY:
Inclusion Criteria:

* All patient with type 2 diabetes with one of the following treatment ongoing : 1) Sulfonylurea 2) Sulfonylurea + OHA. In such patients, if investigator feels that addition of acarbose would be benficial for the patients

Exclusion Criteria:

* According to local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 4564 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Data collection on body weight | 16 weeks
Data collection on blood glucose | 16 weeks
Data collection on Hba1c | 16 weeks
Data collection on pre treatment concomitant diseases | 16 weeks

SECONDARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, India